CLINICAL TRIAL: NCT00528918
Title: Comparison of Apidra to Regular Insulin in Hospitalized Patients
Acronym: Apidra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Meyer - 012
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus, Type II
Keywords: diabetes; hyperglycemia; insulin; Apidra; Glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia; Insulin Resistance | interventions — insulin glulisine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apidra (Active Comparator): Direct 1:1 comparison of Apidra and Regular insulin.
  Interventions: Drug: Glulisine (Apidra)
- Regular (Active Comparator): Direct 1:1 comparison of Apidra and Regular insulin.
  Interventions: Drug: Glulisine (Apidra)

INTERVENTIONS:
Drug: Glulisine (Apidra) — An algorithm to determine the initial doses of insulin and dose adjustments is as follows: Lean subjects (BMI less than 25 kg/m2) will initially receive a total of 0.4 units/kg/day, overweight subjects (BMI 25-30 kg/m2) 0.5 units/kg/day and obese subjects (BMI greater than 30 kg/m2) 0.6 units/kg/day. Fifty percent of the total amount of insulin will be given as Glargine and 50% as regular insulin or Apidra. Supplemental short-acting insulin will be given for hyperglycemia before meals. Automated order sets shall be generated to minimize errors in order entries. Glucose concentrations will be measured before each meal and at bedtime, and if symptomatic. In addition, eight-point blood glucose profiles will be obtained every three days starting on day 2. Dose adjustments will be made to keep blood glucose concentrations between 80 and 120 mg/dl pre-prandially and less than180 mg/dl after meals.

SUMMARY:
The purpose of this study is to compare Apidra (a rapid acting insulin analogue) with Regular insulin (fast acting) in addition to the use of long acting insulin Glargine in hospitalized patients in terms of efficacy and safety in blood glucose control and frequency of low blood glucose. Blood glucose control along with incidence and rate of low blood glucose during the hospitalization shall be of primary interest; length of hospital stay comparing the short acting insulin used shall be the secondary interest.

DETAILED DESCRIPTION:
OBJECTIVES: To compare the rapid acting insulin analogue Apidra with regular insulin in addition to insulin Glargine in hospitalized patients in terms of efficacy and safety, namely Glycemic control and frequency of hypoglycemia. Glycemic control, and incidence and rate of hypoglycemia during the hospitalization shall be the primary endpoints; length of hospital stay according to the short acting insulin used shall be the secondary endpoint.

RESEARCH DESIGN: Randomized, prospective study.

METHODS: Inpatient single center study, planning to enroll 600 patients with type II diabetes admitted to medical or surgical non-ICU service for three days or longer. Subjects will be randomized to Apidra or regular insulin in a 1:1 fashion. Insulin Glargine will be given once a day for basal insulin in all subjects. An algorithm to determine the initial doses of insulin and dose adjustments is as follows: Lean subjects (BMI less than 25 kg/m2) will initially receive a total of 0.4 units/kg/day, overweight subjects (BMI 25-30 kg/m2) 0.5 units/kg/day and obese subjects (BMI greater than 30 kg/m2) 0.6 units/kg/day. Fifty percent of the total amount of insulin will be given as Glargine and 50% as regular insulin or Apidra. Supplemental short-acting insulin will be given for hyperglycemia before meals. Automated order sets shall be generated to minimize errors in order entries. Glucose concentrations will be measured before each meal and at bedtime, and if symptomatic. In addition, eight-point blood glucose profiles will be obtained every three days starting on day 2. Dose adjustments will be made to keep blood glucose concentrations between 80 and 120 mg/dl pre-prandially and less than180 mg/dl after meals. In addition, HbA1c, lipid profile and a fasting plasma C-peptide will be obtained. Two days prior to the anticipated discharge, another HbA1c will be done.

The incidence and the rate of hypoglycemia in each category shall be determined. During the hospitalization, the average of blood glucose measurements at each time point of an 8-point blood glucose profile will be compared; after the hospitalization the HbA1c shall be used. Glycemic control will be compared between groups using ANCOVA adjusting for baseline HbA1c. Hypoglycemic events will be compared between groups using logistic or Poisson regression; length of stay will be compared between groups using survival analysis or the Mann Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be admitted to non-critical care units with expected length of stay of at least three days.
* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Subjects may be of either sex. Female subjects of child-bearing potential must be non-lactating and have a negative pregnancy test before starting the study.
* Subjects must be diagnosed with T2DM or develop hyperglycemia (BG >180 mg/dl) during hospitalization.

Exclusion Criteria:

* Subjects must not be admitted for 'observation' or for expected length of stay of less than three days.
* Subjects must not have Type 1 Diabetes.
* Subjects must not be using rapid acting insulin analogues.
* Subjects must not be receiving nutrition via tube feedings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic events | up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — Carl T. Hayden VA Medical Center
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Meyer C, Boron A, Plummer E, Voltchenok M, Vedda R. Glulisine versus human regular insulin in combination with glargine in noncritically ill hospitalized patients with type 2 diabetes: a randomized double-blind study. Diabetes Care. 2010 Dec;33(12):2496-501. doi: 10.2337/dc10-0957. Epub 2010 Aug 30. PMID 20805258